CLINICAL TRIAL: NCT05320328
Title: SAFETY AND EFFICACY OF INTRA DUCTAL RADIO FREQUENCY ABLATION IN UNRESECTABLE MALIGNANT BILIARY OBSTRUCTION: PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: RADIO FREQUENCY ABLATION IN UNRESECTABLE MALIGNANT BILIARY OBSTRUCTION
Acronym: MBOP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Doctor, Asian Institute of Gastroenterology, India
Other Study IDs: RFA
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Bile Duct Neoplasms; Gall Bladder Carcinoma
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: The study group (A) will receive radio frequency ablation followed by uncovered Self expandable metal stent/Plastic stent placement (one or more)at same procedure.
  Interventions: Device: Radio frequency ablation
- 2: The control group (B) will receive uncovered Self expandable metal stent / Plastic stent (one or more) placement.

INTERVENTIONS:
Device: Radio frequency ablation — Radiofrequency ablation (RFA) uses heat to kill cancer cells. High-frequency electrical currents are passed through a special needle or probe called a needle electrode. The electrical current from the probe heats a small area containing cancer cells to high temperatures, killing the cancer cells. The area around the tumour is also usually treated because it may contain cancer cells.
  Other Names: RFA
  Groups: 1

SUMMARY:
Endoscopic retrograde cholangio pancreatography procedure will performed as per local standard procedure.After common bile duct cannulation,cholangiography will be performed (to confirm the stricture) followed by biliary sphincterotomy. All biliary strictures(Bismuth Type I/II/III/IV) will be enrolled for the study.

Patient opting for Uncovered self expandable metallic stent / Plastic stent will undergo biliary stent placement and considered under control arm Patient opting for radio frequency ablation + Uncovered SEMS/Plastic stent will undergo radio frequency ablation and biliary stent placement and considered under Study arm The RFA probe will be inserted into the bile duct alongwith the guidewire. Keeping the electrode overlapping the stricture, RFA will be performed using a power of 10W for 120 seconds. The electrode will be kept at the ablation site for an additional 1 minute to allow the RFA probe to cool before removal to prevent thermal injury of normal tissue and/or endoscope accessory channel. If the stricture is more than 3 cm, step-by-step RFA will be performed from the superior to inferior aspect. After RFA application, an uncovered SEMS/Plastic stent will be placed.

DETAILED DESCRIPTION:
Placement of self expandable metallic stent is the standard of care in the palliative management of patients with malignant biliary strictures . Relieves biliary obstruction and jaundice.

Self expandable metallic stent provide efficient drainage and have superior patency rates compared with the plastic stents Endoscopic radio frequency ablation combined with stent placement can significantly prolong survival and the stent patency period without increasing the incidence of adverse events in patients with extra hepatic cholangiocarcinoma patient.

Compared to plastic/ metal stent placement alone the addition of radio frequency ablation to stent placement would have better outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. Malignant biliary obstruction confirmed using computed tomography (CT) or abdominal magnetic resonance imaging(MRI), with pathological confirmation whenever possible;
3. Clinical jaundice, a serum bilirubin level greater than 5 mg/dL, and/or cholangitis;
4. ECOG performance status score≤2
5. Un resectability or refusal to be surgically treated.
6. Eligible patients were those with biliary obstruction due to cancer of the gallbladder, or bile ducts; who were considered unsuitable for surgery because of distant metastases, vascular invasion, or severe disability due to age or associated diseases.
7. Non-resectability was established through the consensus opinion of a multidisciplinary tumor board.
8. Written informed consent signed by the patient.

Exclusion Criteria:

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 Subjects
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Prospectively evaluate the safety and efficacy of combining intraductal Radio frequency ablation with biliary metal/ plastic stent placement for patients with malignant biliary obstruction. | 12 months
  satety of radio frequency ablation assessed by complications/adverse effects post procedure and efficacy of the procedure will be assessed by stent patency at the end of one month

SECONDARY OUTCOMES:
Stent patency at 1 year | 12 months
  Stent patency will be estimated by bio chemical parameters (Total bilirubin, Alkaline phosphatase) or ultra sound abdomen scan

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jagtap N, Kumar CS, Lakhtakia S, Ramchandani M, Memon SF, Asif S, Kalapala R, Nabi Z, Basha J, Gupta R, Tandan M, Reddy DN. Adjuvant endobiliary radio-frequency ablation combined with self-expandable biliary metal stents for unresectable malignant hilar strictures: A pragmatic comparative study. Indian J Gastroenterol. 2025 Feb;44(1):72-79. doi: 10.1007/s12664-024-01668-1. Epub 2024 Sep 6. PMID 39240508